CLINICAL TRIAL: NCT05476783
Title: A Multi-center Open-label Long Term Extension Study to Assess the Safety of TB006 in Patients Who Have Completed Protocol TB006AD2102 and in De Novo Patients With Alzheimer's Disease
Brief Title: A Long Term Extension Study to Assess the Safety of TB006 in Participants With Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Resource Constraints
Sponsor: TrueBinding, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB006AD2104
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Open-label Extension; TB006; TB006AD2102; De Novo
MeSH Terms: conditions — Alzheimer Disease | interventions — TB006

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TB006 4000 mg (Experimental): TB006 4000 milligram (mg) via a 1-hour continuous intravenous (IV) infusion will be administered once every 28 day
  Interventions: Drug: TB006

INTERVENTIONS:
Drug: TB006 — Clear to slightly opalescent, sterile solution for injection

SUMMARY:
This is an open-label long term extension study for participants with Alzheimer's disease (AD) who have completed Protocol TB006AD2102 (lead-in study) or participants who would have been eligible for the lead-in study but were not enrolled (de novo). The study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of TB006. The total study duration for each participant will be up to 113 weeks.

DETAILED DESCRIPTION:
The total study duration for each participant will be up to 113 weeks [This includes 101 weeks (2 years) of dosing and a 12-week safety follow-up period]. The number of participants enrolled from the lead-in study will be 100 to 120 and additionally, up to 50 de novo participants, identified by the sponsor, may be included. A total of approximately 150 to 180 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Lead-in study participants are eligible to be included in the study only if they meet the following criteria:

* Completed lead-in Protocol TB006AD2102 (Participants from both study drug and placebo groups) or are eligible for the lead-in study but were not enrolled (de novo).
* Eligibility must be reconfirmed by the investigator for participants who have a gap of more than 28 days between lead-in Protocol TB006AD2102 completion and enrolment in the current study. These participants will undergo the screening procedures in the current Open-label extension (OLE) protocol, with the exception of imaging.
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Females must be of non-childbearing potential.
* Participants or caregiver has the ability to understand the purpose and risks of the study and provide signed and dated informed consent. Participants whose caregiver signs the informed consent must provide their assent.
* Either currently or previously (in pre-AD condition) literate and capable of reading, writing, and communicating effectively with others.
* Participants, along with the caregiver, will be compliant with study visits, procedure.

De novo participants, identified by the sponsor and referred to a participating site, are eligible to be included in the study only if all of the following criteria apply:

* Male and/or female > 50 years of age at the time of signing the informed consent.
* Body weight of ≥ 50 kilograms (kg) and body mass index (BMI) between 18 and 35 kilograms per square meter (kg/m^2), inclusive.
* MMSE score of 24 or less.
* Must be ambulatory.
* Clinical diagnosis of AD consistent with the following:

  1. Probable AD, according to National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA).
  2. Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) - Criteria for Major Neurocognitive Disorder (previously dementia).
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Females must be of non-childbearing potential.
* Participants or caregiver has the ability to understand the purpose and risks of the study and provide signed and dated informed consent. Participants whose caregiver signs the informed consent must provide their assent.
* Either currently or previously (in pre-AD condition) literate and capable of reading, writing, and communicating effectively with others.

Exclusion Criteria:

Lead-in study participants are excluded from the study if any of the following criteria apply:

* Development of an intolerable adverse event or an adverse event that was considered an important safety risk in Protocol TB006AD2102
* Any of the following emerging medical or psychiatric exclusion criteria as defined in the lead-in Protocol TB006AD2102:

  1. Any medical or neurological condition other than AD that in the opinion of the investigator could be a contributing cause of the Participant's dementia
  2. History within the past 6 months or evidence of clinically significant psychiatric illness like major depression, schizophrenia, or bipolar affective disorder
  3. Diagnosis of a dementia-related central nervous system (CNS) disease other than AD (eg, Parkinson's Disease, Huntington's Disease, frontotemporal dementia, multi-infarct dementia, dementia with Lewy bodies, or normal pressure hydrocephalus).
  4. Identification of other known cause of dementia or any other clinically significant contributing co-morbid pathologies at screening MRI
  5. Any contraindications to having a brain MRI eg, pacemaker; non-MRI compatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia)
  6. Any untreated or unstable clinically significant medical condition like hypertension, diabetes, chronic obstructive pulmonary disorder, asthma, or depression
  7. Any clinically significant findings in medical examination, including physical examination, 12-lead electrocardiogram (ECG), clinical laboratory tests.
  8. Undergone major surgery <= 2 months before study drug administration.
  9. Loss of more than 100 milliliters (mL) blood (eg, a blood donation) within 2 months before first study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months before Day 1, or plans to donate blood during the study or within 3 months after the study.
  10. Regular alcohol consumption within 6 months prior to the study defined as: an average weekly (QW) intake of > 20 units for males or > 16 units for females. One unit is equivalent to 8 grams (g) of alcohol.
  11. Meets DSM-5 criteria for moderate or severe substance use disorder within the past 12 months, or has a positive test for substances of abuse, or has used substances, including but not limited to opiates, methadone, buprenorphine, methamphetamine, cocaine, amphetamines recreationally within the past 12 months.
  12. Unable to complete this study for other reasons or the investigator believes the Participant should be excluded.
* Since participating in Protocol TB006AD2102, the participant has participated in another drug, biologic, device, or a clinical study or treatment with an investigational drug or approved therapy for investigational use.
* Any clinically significant findings in medical examination. This includes physical examination, 12-lead ECG, or clinical laboratory tests on the final visit in Protocol TB006AD2102 or on the Baseline visit in this study. Participants who are coronavirus disease of 2019 (COVID-19)-positive at Screening (or end of treatment [EOT] from lead-in study) must delay the start of the study until they are COVID-19-negative. They may be retested at weekly intervals.
* Participants who have undergone major surgery since enrolment in Protocol TB006AD2102 will be considered on a case-by-basis.

De Novo participants are excluded from the study if any of the following criteria apply:

* Any medical or neurological condition other than AD that in the opinion of the investigator could be a contributing cause of the participant's dementia
* History within the past 6 months or evidence of clinically significant psychiatric illness (eg, major depression, schizophrenia, or bipolar affective disorder).
* Diagnosis of a dementia-related CNS disease other than AD (eg, Parkinson's Disease, Huntington's Disease, frontotemporal dementia, multi-infarct dementia, dementia with Lewy bodies, normal pressure hydrocephalus).
* Identification of other known cause of dementia or any other clinically significant contributing co-morbid pathologies at screening MRI, in the opinion of the investigator.
* Participation in any other drug, biologic, device, or clinical study or treatment with any investigational drug or approved therapy for investigational use within 30 days (or 5 half-lives, whichever is longer) prior to screening, and/or participation in any other clinical study involving experimental medications for AD within the 60 days (or 5 half-lives, whichever is longer) prior to screening.
* Any contraindications to having a brain MRI eg, pacemaker; non-MRI-compatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia).
* Any untreated or unstable clinically significant medical condition (ie, hypertension, diabetes, chronic obstructive pulmonary disorder, asthma, depression, etc.) as judged by the investigator.
* Any clinically significant findings in medical examination, including physical examination, 12-lead ECG, clinical laboratory tests.
* Undergone major surgery <= 2 months before study drug administration.
* Loss of more than 100 mL blood (eg, a blood donation) within 2 months before first study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months before Day 1, or plans to donate blood during the study or within 3 months after the study.
* Recent (3-month) history of a positive COVID-19 test result or disease symptoms of COVID-19 disease such as shortness of breath, cough, rhinorrhea, and sore throat, etc.
* Known history of, or a positive test result for Hepatitis B surface antigen (HBsAg), immunoglobulin M antibody to Hepatitis B core antigen (IgM anti HBc), anti-hepatitis C virus antibodies (HCV), or human immunodeficiency virus (HIV) types 1 or 2 at screening. Participants with a documented history of treatment for Hepatitis C are otherwise eligible to participate.
* Regular alcohol consumption within 6 months prior to the study defined as: an average QW intake of > 20 units for males or > 16 units for females.
* Meets DSM-5 criteria for moderate or severe substance use disorder within the past 12 months, or has a positive test for substances of abuse, or has used substances, including but not limited to opiates, methadone, buprenorphine, methamphetamine, cocaine, amphetamines recreationally within the past 12 months.
* Unable to complete this study for other reasons or the investigator believes that he or she should be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 113 weeks
Number of participants with Clinically Significant Clinical Laboratory Parameter Values | Up to 113 weeks
Number of Participants with Clinically Significant Vital Sign Values | Up to 113 weeks
Number of Participants with Clinically Significant 12-Lead electrocardiogram Findings | Up to 113 weeks
Change from Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline and up to 113 weeks
  The C-SSRS is a suicidal ideation and behavior rating scale with yes/no responses. For each of the 5 items of the C-SSRS related to suicidal ideation intensity, an individual's degree of suicidal ideation is rated on a 0-5 scale with 0: no suicidal behavior and 5: active suicidal ideation. The total score is the sum of the 5 intensity item scores (total score ranges from 0 to 25). Higher scores in the scale indicate greater disease severity.
Number of Participants with Clinically Significant Physical Examination Findings | Up to 113 weeks
Number of Participants with Clinically Significant Neurological Examination Findings | Up to 113 weeks
Number of participants with magnetic resonance imaging (MRI) abnormalities | Up to 113 weeks
Plasma concentration of TB006 | Pre-dose, and Weeks 1, 5, 9, 13, 17, 21, 25, 45, 73, 101 and 113
Number of Participants with Anti-TB006 Antibodies | Up to 113 weeks

SECONDARY OUTCOMES:
Change from Baseline in Clinical Dementia Rating Scale-Sum of Boxes (CDR SB) score | Baseline and up to Week 101
  The CDR scale is a clinician-rated dementia staging system that tracks the progression of cognitive impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care). Each category is scored on a 5-point scale in which None = 0, Questionable = 0.5, Mild = 1, Moderate = 2, and Severe = 3. The global CDR score is established by clinical scoring rules and has values of 0 (no dementia), 0.5, (questionable dementia), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia). The Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) is obtained by adding the ratings in each of the 6 categories and ranges from 0 to 18 with higher scores indicative of greater impairment.
Change from Baseline in cognitive functioning | Baseline and up to Week 101
  Cognitive functioning will be measured by Cognitive Drug Research system (CDR) Computerized Assessment system. It assesses different cognitive domains: attention, working memory, episodic memory, and executive function. It contains 11 tests and is performed on a tablet-like device. Participants respond via 'Yes (1)' and 'No (0)' buttons on a two-button response box. The minimum possible score is 0 and maximum possible score is 11. Higher score indicates better cognitive function
Change from Baseline in Mini Mental State Examination (MMSE) score | Baseline and up to Week 101
  Global cognitive functioning is measured by MMSE. MMSE is a neuropsychological test for the evaluation of intellectual efficiency disorders and the presence of cognitive impairment. The total score is between a minimum of 0 (worse cognitive function) and a maximum of 30 points (normal cognitive function). A lower score indicates severe impairment of cognitive abilities and a higher score indicates cognitive normality.
Change from Baseline in Neuropsychiatry Inventory (NPI) score | Baseline and up to Week 101
  The NPI is a condition-specific measure designed to assess 12 behavioral disturbances, namely delusions, hallucinations, depression/dysphoria, anxiety, agitation/aggression, elation/euphoria, disinhibition, irritability/lability, apathy, aberrant motor activity, night-time behavior disturbances, and appetite/eating abnormalities. The frequency is scored from 0 (never) to 4 (very frequently) and severity ranges between 0 (none) to 3 (marked). The domain score is obtained by multiplying frequency and severity scores. The total NPI score is the sum total of all individual domain scores (0-144). A higher score indicates abnormal behaviour.
Change from Baseline in EuroQol 5 Dimension 5-Level quality of life (EQ 5D 5L QoL) total score | Baseline and up to Week 101
  EuroQol 5 is a self-reported description of participant's current health in 5 dimensions i.e., mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants to grade their own current level of function in each dimension into one of three degrees of disability (severe, moderate or none). Score ranges between 1 (no problem) and 3 (significant problem). higher scores indicating higher health utility. The total score is the sum total of all individual domain scores (5-15). Higher scores indicates poor quality of life.
Change from Baseline in brain atrophy measured by MRI | Baseline and up to Week 113
Change from Baseline in amyloid plaque using positron emission tomography (PET) imaging | Baseline and up to Week 113
Change from Baseline in brain volume using MRI | Baseline and up to Week 113

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Delray Beach, Florida
  - Clinical Trial Site, Lady Lake, Florida
  - Clinical Trial Site, Maitland, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Winter Park, Florida
  - Clinical Trial Site, Decatur, Georgia
  - Clinical Trial Site, Matthews, North Carolina
  - Clinical Trial Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No